CLINICAL TRIAL: NCT04395287
Title: Prospective Associations Between Screen Media Use and Physical Activity in Preschool Children: Findings From the Motor Skills in PreSchool (MIPS) Study
Brief Title: Prospective Associations Between Screen Media Use and Physical Activity in Preschool Children
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: European Research Council (Other); University of Sydney (Other)
Responsible Party: Sponsor
Other Study IDs: S-2015-0178; 2015-57-0008 (Other: Danish Data Protection Agency)
Record Dates: First submitted 2020-04-28; First posted 2020-05-20 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Screen Time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preschool children: Attending public preschools in Svendborg, Denmark, at the time of recruitment
  Interventions: Behavioral: Leisure screen time

INTERVENTIONS:
Behavioral: Leisure screen time — Questionnaire-based assessment of typical amount of time per week spent using screen-based media devices during leisure, assessed at two time points. Continuously scaled in main analyses; a difference is computed (18-month follow-up value minus baseline value). Additionally, screen time amount at the two time points will be scaled categorically, according to being classified as low or high according to WHO criteria for preschool children (Low (recommended): <=1 hour/day, high: >1 hour/day): High-high, high-low, low-high, and low-low.

SUMMARY:
The aims of this study are as follows:

* The primary aim is to investigate the relationship between changes in screen media use with changes in non-sedentary time (time, min/day, spent in activities other than lying and sitting) during leisure (outside nursery) from baseline to 18-month follow-up.
* The secondary aim is to investigate the relationship between changes in screen media use and time (min/day) spent in specific daily activities (lying, sitting, moving, standing, walking, and running) and changes in moderate-to-vigorous intensity physical activity during leisure.

DETAILED DESCRIPTION:
The current study is a secondary, observational investigation of data from The Motor Skills in PreSchool (MIPS) study. The MIPS study was initiated in 2016 and included preschool children (3-6 years of age) attending public preschools in the Municipality of Svendborg, in Denmark. A subset of the preschools included an intervention component, whose aim was optimization of motor skills. In this study, the children's screen media use was assessed via questionnaire and physical activity was assessed using two Axivity AX3 (Axivity Ltd., Newcastle upon Tyne, United Kingdom) triaxial accelerometers - one placed at the hip and one at the lower back - at both baseline and at 18-month follow-up. Time spent in distinct activity types (sitting, moving, standing, biking, running, walking, and lying down) are determined from the acceleration measured with the thigh worn device. In addition, data on relevant covariates was also collected. Having data on both exposure and outcome at baseline and follow-up renders detailed longitudinal assessments possible. Furthermore, daily schedule (proxy based on reporting by parents and pedagogical personnel) information on the children introduces the possibility of domain-specific analyses of physical activity, as we can time annotate the data into different sections of the children's daily routine.

ELIGIBILITY:
Inclusion:

- All children who at the time of recruitment attended public preschools in the Municipality of Svendborg

Exclusion:

- None

Ages: 3 Years to 6 Years | Sex: All
Age Groups: Child
Study Population: 3-6-year-old children attending public preschools in Municipality of Svendborg at the time of recruitment (fall of 2016), and their parents
Sampling Method: Probability Sample
Enrollment: 887 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Non-sedentary time during leisure | 18 months
  Change in mean min/day

SECONDARY OUTCOMES:
Time spent lying down during leisure | 18 months
  Change in mean min/day
Time spent sitting during leisure | 18 months
  Change in mean min/day
Time spent 'moving' during leisure | 18 months
  Change in mean min/day of standing activity with a small degree of bodily movement
Time spent standing during leisure | 18 months
  Change in mean min/day
Time spent walking during leisure | 18 months
  Change in mean min/day
Time spent running during leisure | 18 months
  Change in mean min/day

CONTACTS AND LOCATIONS:
Overall Officials: Line G. Olesen, Ph.D., Principal Investigator — University of Southern Denmark
Locations (1):
- Research in Childhood Health Research Center, Odense, Southern Danmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hestbaek L, Andersen ST, Skovgaard T, Olesen LG, Elmose M, Bleses D, Andersen SC, Lauridsen HH. Influence of motor skills training on children's development evaluated in the Motor skills in PreSchool (MiPS) study-DK: study protocol for a randomized controlled trial, nested in a cohort study. Trials. 2017 Aug 29;18(1):400. doi: 10.1186/s13063-017-2143-9. PMID 28851412

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/87/NCT04395287/SAP_000.pdf